CLINICAL TRIAL: NCT06581159
Title: Phase 1b Double-Blind, Placebo-Controlled, MAD Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS135 in Obese Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction
Brief Title: Study of HS135 in Obese Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: 35Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS135-003
Record Dates: First submitted 2024-08-09; First posted 2024-09-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind, Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): HS135 Subcutaneous Injection
  Interventions: Biological: HS135
- Placebo (Placebo Comparator): Subcutaneous Injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HS135 — Subcutaneous Injection
  Arms: Investigational Product
Other: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
A Study of HS135 for the Treatment of in Obese Patients with Pulmonary Hypertension and Heart Failure with Preserved Ejection Fraction (PH-HFpEF)

DETAILED DESCRIPTION:
Phase 1b, Multicenter, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS135 in Obese Patients with Pulmonary Hypertension and Heart Failure with Preserved Ejection Fraction

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet at least all the following criteria:

1. Male or female, >18 years of age.
2. CardioMEMS™ Heart Failure System implanted during standard of care at least 90 days before Screening.
3. Established diagnosis of HFpEF with Left Ventricular Ejection Fraction (LVEF) at least 45% as measured by echocardiography during Screening.
4. New York Heart Association (NYHA) class II, III or IV heart failure symptoms.
5. BMI ≥ 30 kg/m2.
6. Ability to adhere to study visit schedule and understand and comply with all protocol requirements.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Decompensated heart failure.
2. Admission for an acute coronary syndrome, percutaneous coronary intervention, or cardiac surgery within 30 days prior to Screening.
3. Implantation of cardiac resynchronization therapy (CRT) device within 90 days prior to Screening.
4. Planned cardiovascular revascularization or major cardiac surgery or planned implantation of CRT device.
5. History of heart transplant or on heart transplant list.
6. Uncontrolled systemic hypertension.
7. Patients who have an abnormality in echocardiography or electrocardiogram that in the opinion of the investigator increases the risk of participating in the study.
8. Patients who have full pneumonectomy or a severe chronic pulmonary disorder that in the opinion of the investigator increases the risk of participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence and Number of Adverse Events (AEs) | Up to 24 weeks
  An AE is any untoward medical occurrence in a patient or clinical trial patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The incidence and number of patients who experience an AE will be reported.
Change from Baseline in Clinical Laboratory Parameters (Hematology): White Blood Cell Count | Up to 24 weeks
  Blood samples will be collected to determine the White Blood Cell Count at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Hematology): Platelet Count | Up to 24 weeks
  Blood samples will be collected to determine the Platelet Count at designated time points up to 24 weeks.
Change from Baseline in Clinical Laboratory Parameters (Hematology): Red Blood Cell Count | Up to 24 weeks
  Blood samples will be collected to determine the Red Blood Cell Count at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Hematology): Hemoglobin | Up to 24 weeks
  Blood samples will be collected to determine concentration of Hemoglobin at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Hematology): Hematocrit | Up to 24 weeks
  Blood samples will be collected to determine concentration of Hematocrit at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Albumin | Up to 24 weeks
  Blood samples will be collected to determine concentration of Albumin at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Aspartate aminotransferase (AST) | Up to 24 weeks
  Blood samples will be collected to determine concentration of AST designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Alanine aminotransferase (ALT) | Up to 24 weeks
  Blood samples will be collected to determine concentration of ALT designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Alkaline phosphatase (ALP) | Up to 24 weeks
  Blood samples will be collected to determine concentration of ALP designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Total Bilirubin | Up to 24 weeks
  Blood samples will be collected to determine concentration of Total Bilirubin at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Calcium | Up to 24 weeks
  Blood samples will be collected to determine concentration of Calcium at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Creatinine | Up to 24 weeks
  Blood samples will be collected to determine concentration of Creatinine at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Glucose | Up to 24 weeks
  Blood samples will be collected to determine concentration of Glucose at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Urea | Up to 24 weeks
  Blood samples will be collected to determine concentration of Urea at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Total Cholesterol | Up to 24 weeks
  Blood samples will be collected to determine concentration of Total Cholesterol at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): High-density Lipoprotein-cholesterol (HDL-c) | Up to 24 weeks
  Blood samples will be collected to determine concentration of HDL-c at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Low-density Lipoprotein-cholesterol (LDL-c) | Up to 24 weeks
  Blood samples will be collected to determine concentration of LDL-c at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Chloride | Up to 24 weeks
  Blood samples will be collected to determine concentration of Chloride at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Potassium | Up to 24 weeks
  Blood samples will be collected to determine concentration of Potassium at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Biochemistry): Sodium | Up to 24 weeks
  Blood samples will be collected to determine concentration of Sodium at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Blood (occult) | Up to 24 weeks
  Urine samples will be collected to determine the presence of Blood (occult) at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Ketones | Up to 24 weeks
  Urine samples will be collected to determine the presence of Ketones at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Leukocyte Esterase | Up to 24 weeks
  Urine samples will be collected to determine the presence Leukocyte Esterase of at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Nitrites | Up to 24 weeks
  Urine samples will be collected to determine the presence of Nitrites at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Bilirubin | Up to 24 weeks
  Urine samples will be collected to determine the presence of Bilirubin at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Glucose | Up to 24 weeks
  Urine samples will be collected to determine the presence of Glucose at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Urobilinogen | Up to 24 weeks
  Urine samples will be collected to determine concentration of Urobilinogen at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Protein | Up to 24 weeks
  Urine samples will be collected to determine the presence of Protein at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): pH | Up to 24 weeks
  Urine samples will be collected to determine the pH at designated time points up to 24 weeks
Change from Baseline in Clinical Laboratory Parameters (Urinalysis): Specific Gravity | Up to 24 weeks
  Urine samples will be collected to determine the Specific Gravity at designated time points up to 24 weeks

SECONDARY OUTCOMES:
Change from Baseline in mean pulmonary artery diastolic pressure (mPADP) at designated time points up to 24 weeks | Up to 24 weeks
  To determine mean pulmonary artery diastolic pressure (mPADP)
Change from Baseline in mean pulmonary artery pressure (mPAP) at designated time points up to 24 weeks | Up to 24 weeks
  To determine mean pulmonary artery pressure (mPAP)
Change from Baseline in mean pulmonary artery systolic pressure (mPASP) at designated time points up to 24 weeks | Up to 24 weeks
  To determine mean pulmonary artery systolic pressure (mPASP)
Change in New York Heart Association (NYHA) Class at designated time points up to 24 weeks | Up to 24 weeks
  To determine change in New York Heart Association (NYHA) Class at Week 24
Change from Baseline in number of hospitalizations or urgent outpatient visits for heart failure during the treatment period at designated time points at designated time points up to 24 weeks | Up to 24 weeks
  To determine number of hospitalizations or urgent outpatient visits for heart failure during the treatment period
Change from Baseline to Week 24 in N-terminal pro-B-type natriuretic peptide (NT-proBNP) at designated time points up to 24 weeks | Up to 24 weeks
  To determine N-terminal pro-B-type natriuretic peptide (NT-proBNP)
Change from Baseline in 6-minute walk distance (6MWD) at designated time points up to 24 weeks | Up to 24 weeks
  To determine 6-minute walk distance (6MWD)
Change from Baseline in Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CS) and Kansas City Cardiomyopathy Questionnaire-Overall Summary Score (KCCQ-OS) at designated time points up to 24 weeks | Up to 24 weeks
  To determine change from Baseline in Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CS) and Kansas City Cardiomyopathy Questionnaire-Overall Summary Score (KCCQ-OS) at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Champagne, M.Sc., Study Director — 35Pharma Inc
Locations (2):
- United States (2):
  - Site-104, Phoenix, Arizona
  - Site-105, Kansas City, Missouri